CLINICAL TRIAL: NCT01401283
Title: Multi-center, Prospective, Randomized Outcome Study Comparing Continuous Cardiac Index Trending Via a Radial Arterial Line Versus Standard Care in General Surgical Patients
Brief Title: GDT by Cardiac Index Trending Via a Radial Arterial Line in General Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Collaborators: Northern State Medical University (Other); Szeged University (Other); University of Kiel (Other); University of Witten/Herdecke (Other); University of Valencia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 797726
Record Dates: First submitted 2011-07-08; First posted 2011-07-25 (Estimated); Results first posted 2016-02-05 (Estimated); Last update posted 2016-02-05 (Estimated); Status verified 2016-01

CONDITIONS: Reduction of Length of Hospitality Stay, Reduction of Perioperative Complications

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Study group (Active Comparator): intraoperative guidance of hemodynamics by measures of cardiac index and pulse pressure variation, measurement of cardiac output and pulse pressure variation, hemodynamic optimization according to cardiac index and pulse pressure variation
  Interventions: Device: measurement of cardiac output and pulse pressure variation
- Control group (No Intervention): hemodynamic management according to institutional clinical standards

INTERVENTIONS:
Device: measurement of cardiac output and pulse pressure variation — hemodynamic optimization according to cardiac index and pulse pressure variation
  Arms: Study group

SUMMARY:
This is a multi-Center, prospective, randomized Outcome Study comparing continuous cardiac index trending via a radial arterial line versus standard care in general surgical patients

DETAILED DESCRIPTION:
This is a multi-Center, prospective, randomized Outcome Study comparing continuous cardiac index trending via a radial arterial line versus standard care in general surgical patients Clinical outcome of patients undergoing major abdominal surgery is explored in two different groups. In one group hemodynamic management is guided by the internal standard of the anesthesiological department. In the other group fluid management is goal directed by by continuous cardiac index trending via a radial arterial line and pulse pressure variation.

ELIGIBILITY:
Inclusion Criteria:

* major abdominal surgery
* duration of surgery > 2 hours

Exclusion Criteria:

* age < 18 years
* scheduled postoperative icu treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2011-07; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel A Reuter, MD, Principal Investigator — Universitätsklinikum Hamburg-Eppendorf
Locations (1):
- University Medical Center Hamburg-Eppendorf, Hamburg, Germany

REFERENCES:
- [Derived] Salzwedel C, Puig J, Carstens A, Bein B, Molnar Z, Kiss K, Hussain A, Belda J, Kirov MY, Sakka SG, Reuter DA. Perioperative goal-directed hemodynamic therapy based on radial arterial pulse pressure variation and continuous cardiac index trending reduces postoperative complications after major abdominal surgery: a multi-center, prospective, randomized study. Crit Care. 2013 Sep 8;17(5):R191. doi: 10.1186/cc12885. PMID 24010849

RESULTS

PARTICIPANT FLOW:
Groups:
- Study Group: intraoperative guidance of hemodynamics by measures of cardiac index and pulse pressure variation
  measurement of cardiac output and pulse pressure variation: hemodynamic optimization according to cardiac index and pulse pressure variation
Period: Overall Study
Arm/Group | Study Group | Control Group
Started | 89 | 91
Completed | 79 | 81
Not Completed | 10 | 10
Not completed — surgery cancelled | 5 | 8
Not completed — preoperative arrhythmia | 5 | 0
Not completed — no central venous access | 0 | 1
Not completed — suspicion of malignant hyperthermia | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Study Group | Control Group | Total
Number analyzed (Participants) | 89 | 91 | 180
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 64 | 55 | 119
  >=65 years | 25 | 36 | 61
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37 | 36 | 73
  Male | 52 | 55 | 107
Region of Enrollment [Number; unit: participants]
  Germany | 89 | 91 | 180

OUTCOME MEASURES:

1. Primary Outcome: Postoperative Complications
Description: Categories of postoperative complications: Infection (respiratory, abdominal, UTI, wound), Respiratory (prolonged need for ventilation), Cardiovascular (edema, arrythmia, hypotension, AMI, stroke), Abdominal (constipation), Renal (urine output <500ml/d, ARF)
Time Frame: Participants will be followed from end of surgery for the duration of stay in the recovery room, for the duration of the complete hospital stay, an expected average of ten 10 days
Measure: Number; unit: numbers of complications
Arm/Group | Study Group | Control Group
Number analyzed (Participants) | 89 | 91
numbers of complications | 52 | 72

2. Secondary Outcome: Hospital Stay
Description: length of stay in the postoperative care unit, length of hospital stay
Time Frame: Participants will be followed for the duration of hospital stay, an expected average of 10 days
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Study Group | Control Group
Number analyzed (Participants) | 89 | 91
days | 11 [7 to 15] | 10 [4.1 to 15.9]

ADVERSE EVENTS:
Arm/Group | Study Group | Control Group
Serious Adverse Events (participants affected / at risk) | 0/79 | 0/81
Other Adverse Events (participants affected / at risk) | 0/79 | 0/81

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No